CLINICAL TRIAL: NCT00425035
Title: A Two-part, Multiple Dose Clinical Trial Evaluating the Safety and Effectiveness of ABX-EGF in Patients With Renal Carcinoma
Brief Title: Safety and Efficacy Study of ABX-EGF in Patients With Renal Cancer, Part 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20020374; Abgenix protocol No. ABX-0303; Immunex protocol No. 054.0003; NCT00036530 (obsolete NCT alias)
Record Dates: First submitted 2007-01-18; First posted 2007-01-22 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Advanced Renal Cell Carcinoma
Keywords: Renal Cancer
MeSH Terms: conditions — Kidney Neoplasms | interventions — Panitumumab

INTERVENTIONS:
Drug: Panitumumab (ABX-EGF)

SUMMARY:
Multicenter, 2-part, multiple-dose study designed to evaluate the safety and effectiveness of weekly administration of panitumumab in subjects with renal carcinoma. Part 1 was initiated in 2001 and will not be presented here. Part 2 was designed to examine a dose of 2.5 mg/kg/wk in 2 cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and sign an IRB approved Informed Cosent Form
* Male or female 18 years of age or older
* Female patients who are post menopausal (no menstrual period for a minimum of six months), surgically sterilized, or are using an oral or implanted contraceptive, double barrier birth control, or an IUD and have a negative serum pregnancy test upon entry into this study; or male patients willing to use contraception upon enrollment into this study
* Pathologic diagnosis of renal cell carcinoma by fine needle aspirate or tissue biopsy
* Prior nephrectomy
* Prior Therapy:

  1. Cohort 1 only: Previously received and failed one prior biotherapy, defined as IL-2 therapy or interferon-alpha (alone or in combination); Karnosky score of > or = 70%
  2. Cohort 2 only: No prior therapy except nephrectomy and fall within the Motzer intermediate group with one or two of the risk factors, as defined in teh Study Design section.
* Has bi-dimensionally measurable disease
* Has tumor tissue available for diagnostics (acceptable: biopsy, nephrectomy tissue, fine needle aspirate, or archived tissue that is formalin fixed and paraffin embedded). In cases when a fresh biopsy can be obtained, the biopsy should be divided into two; one half should be formalin fixed, and the other half frozen. Tumor samples must be received at the central laboratory prior to patient regisration.
* Adequate hematologic data, as follows:

  1. ANC > 1.5 x 109/L
  2. Platelet count > 100x 109/L
* Adequate renal function, as follows:

  1. Creatinine < or = 2.2mg/dL
* Adequate hepatic function, as follows:

  1. Alkaline phosphatase < or = 3x ULN
  2. AST < or = 3x ULN
  3. ALT < or = 3x ULN
  4. Total bilirubin < or = 1.5x ULN

Exclusion Criteria:

* Brain metastases
* Cohort 1 only: Hypercalcemia (calcium level outside the upper limit of normal; antihypercalcemic treatment is allowed)
* Cancer therapy within 30 days of ABX-EGF infusion (hormone therapy is allowed; steroid therapy is only allowed if it is replacement therapy)
* Use of any investigational drug within 30 days of ABX-EGF infusion
* Prior treatment with any anti-EGFr agents
* Left ventricular ejection fraction < 45%, as measured by MUGA Scan
* Myocardial infarction within one year prior to entering the study
* Has other cancer that has been active and required treatment within the past 5 years (prior renal cell carcinoma, basal cell carcinoma, or cervical carcinoma in situ are allowed)
* Pregnant or breast feeding female; male or female of childbearing potential (defined as: post menarche and is biologically capable of becoming pregnant) unwilling to use birth control (as defined in the inclusion criteria) during and for 1 month following treatment
* Known to be HIV positive
* History of any chronic medical or psychiatric condition or laboratory abnormality that in the opinion of the Investigator may increase the risks associated with study participation or study drug administration or may interfere with the interpretation of study results
* Allergy to the ingredients of the study medication or to Staphylococcus Protein A

Age Groups: Child, Adult, Older Adult
Enrollment: 115
Dates: Start 2003-02

PRIMARY OUTCOMES:
Part 2, Cohort 1: Efficacy: Tumor response rate (CR or PR) measured at 8 weeks
Part 2, Cohort 1: Safety: Incidence and severity of AEs
Part 2, Cohort 2: Time to disease progression

SECONDARY OUTCOMES:
Part 2, Cohort 1: Time to disease progression
Part 2, Cohorts 1 & 2: Survival time
Part 2, Cohorts 1 & 2: PFS
Part 2, Cohorts 1 & 2: Best overall response rate
Part 2, Cohorts 1 & 2: Tumor response rate at Weeks 15, 23, 31, and 39
Part 2, Cohorts 1 & 2: Duration of response
Part 2, Cohorts 1 & 2: Percent of patients with progressive disease (measured at 8 weeks following initiation of panitumumab treatment)
Part 2, Cohorts 1 & 2: Time to CR
Part 2, Cohorts 1 & 2: Time to response (PR or CR)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Rowinsky EK, Schwartz GH, Gollob JA, Thompson JA, Vogelzang NJ, Figlin R, Bukowski R, Haas N, Lockbaum P, Li YP, Arends R, Foon KA, Schwab G, Dutcher J. Safety, pharmacokinetics, and activity of ABX-EGF, a fully human anti-epidermal growth factor receptor monoclonal antibody in patients with metastatic renal cell cancer. J Clin Oncol. 2004 Aug 1;22(15):3003-15. doi: 10.1200/JCO.2004.11.061. Epub 2004 Jun 21. PMID 15210739
- See also: FDA-approved Drug Labeling — http://www.vectibix.com/
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com